CLINICAL TRIAL: NCT00477659
Title: A Single Center Study To Examine Neural Correlates Of Cognition In Subjects With Mild Alzheimer's Disease After Three Months Of Open Label Donepezil HCl (Aricept® ) Treatment
Brief Title: Neural Correlates In Mild Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-416; A2501055 (Other: Pfizer)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2009-05

CONDITIONS: Alzheimer's Disease
Keywords: Functional magnetic resonance imaging examination; Alzheimer's Disease; Donepezil hydrochloride; Aricept
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Donepezil hydrochloride (Experimental)
  Interventions: Drug: Donepezil hydrochloride

INTERVENTIONS:
Drug: Donepezil hydrochloride — Donepezil hydrochloride 5 mg per day orally, once daily for 4 weeks, followed by 10 mg per day (two 5-mg tablets) for 8 weeks
  Other Names: E2020, Aricept

SUMMARY:
The objective of this study was to identify neural correlates of cognitive improvement after 3 months of donepezil hydrochloride treatment using either or both of two functional magnetic resonance imaging (fMRI) measures - the functional Hippocampus Connectivity Index (HCI) and Cerebral Blood Flow (CBF) Perfusion; in the Medial Temporal Lobe (MTL) network in subjects in the early stage of Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 50 and older with mild Alzheimer's disease (MMSE scores of 20 to 30 are allowed).
* Diagnostic evidence of Alzheimer's disease.
* Previous use of cholinesterase inhibitors (other than Aricept) and memantine allowed.

Exclusion Criteria:

* Prior use of Aricept, pacemakers and insulin dependent diabetes are not allowed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2008-08-15 (Actual); Study Completion 2008-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at one investigative site in the United States from 23 July 2007 to 15 August 2008.
Pre-assignment Details: Out of the 16 participants who were screened, 14 participants were enrolled into the study.
Groups:
- Donepezil Hydrochloride: Participants received donepezil hydrochloride 5 mg per day orally, once daily for 4 weeks, followed by 10 mg per day (two 5-mg tablets) for 8 weeks.
Period: Overall Study
Arm/Group | Donepezil Hydrochloride
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) set included all participants who received at least one dose of study medication, had a baseline efficacy evaluation, and had at least one post-baseline efficacy evaluation.
Groups:
- Donepezil: Participants received donepezil hydrochloride 5 mg per day orally, once daily for 4 weeks, followed by 10 mg per day (two 5-mg tablets) for 8 weeks.
Arm/Group | Donepezil
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 Based on Hippocampus Connectivity Index (HCI)
Description: All neuroimaging procedures were performed on a research-dedicated GE 3.0 Tesla whole-body Excite scanner with 8-channel phase-array head coil. Resting-state functional magnetic resonance imaging (fMRI) of the medial temporal lobe (MTL) was performed. The functional HCI was derived from the MTL network using a data driven approach corresponding voxel time courses from the fMR images were processed to extract low frequency fluctuations. Functional connectivity was quantified by calculating the cross-correlation of each voxel time course in the hippocampus to all voxel time courses of the whole brain and the mean of absolute cross-correlation coefficients between a hippocampus voxel to the whole-brain voxels. HCI was then calculated as the average of all hippocampus cross-correlation coefficients. Change from baseline (CFB) was calculated using the CBF-Perfusion Processing Method. A positive change from baseline for HCI indicates improved function.
Time Frame: Week 12
Population: The ITT set included all participants who received at least one dose of study medication, had a baseline efficacy evaluation, and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 14
percent change | 7.47 (17.23)

2. Secondary Outcome: Change From Baseline at Week 12 in Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS)-Cog Score
Description: The ADAS-cog is a 13-item performance-based test that examines selected aspects of cognition including memory, orientation, attention, reasoning, language, and praxis. Total score ranges from 0 to 70 with higher scores indicating greater cognitive impairment. A decrease from baseline indicates improved cognitive function. The ADAS-cog was administered by a trained individual unaware of adverse events reported during this trial.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 14
score on a scale
  Baseline | 12.0 (4.85)
  Change at Week 12 | -1.6 (2.81)

3. Secondary Outcome: Change From Baseline at Week 12 in Mini-Mental State Examination (MMSE) Score
Description: MMSE was a 11-item scale to measure cognitive status where a higher score indicated better cognitive state. The score ranged from 0 to 30, with a higher score indicating better function. A positive change score indicated improvement from baseline. The mean change was analyzed by Wilcoxon's signed rank test.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 14
score on a scale
  Baseline | 26.1 (1.33)
  Change at Week 12 | 0.1 (2.70)

4. Secondary Outcome: Change From Baseline at Week 12 in the Instrumental Activities of Daily Living (IADL) Assessment Score
Description: IADL Scale measures 7 areas of more complex activities required for optimal independent functioning, as reported by the caregiver. The scoring indicates whether the participant was completely independent (3), requires assistance (2), or is dependent (1) for the performance of each activity. A summary score ranges from 7 (high function, independent) to 21 (low function, dependent). The mean change was analyzed by Wilcoxon's signed rank test. A decrease from Baseline to Week 12 indicates improved function.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 14
score on a scale
  Baseline | 13.1 (3.71)
  Change at Week 12 | -0.3 (2.70)

5. Secondary Outcome: Change From Baseline at Week 12 in the Neuropsychiatric Inventory (NPI) Score
Description: NPI was a 12-item caregiver-based assessment of behavioral disturbances commonly occurring in participants with AD. NPI includes 12 sections which are Delusions, Hallucinations, Agitation, Depression, Anxiety, Euphoria, Apathy, Disinhibition, Irritability, Aberrant motor behavior, Night-time behaviors and Appetite and eating disorders. The score of each section ranges from 0 to 12, and higher score means higher severity and frequency of the neuropsychiatric disturbances. The mean change was analyzed by Wilcoxon's signed rank test.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil Hydrochloride
Number analyzed (Participants) | 14
score on a scale
  Baseline | 9.2 (10.00)
  Change at Week 12 | -3.4 (11.25)

ADVERSE EVENTS:
Time Frame: All adverse events were collected from first dose of study drug (Baseline) up to 30 days after last dose of study drug (approximately up to 12 weeks)
Description: Safety analysis set included all participants who received at least one dose of study medication.
Arm/Group | Donepezil Hydrochloride
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Hydrochloride (N=14)
Decreased appetite (Metabolism and nutrition disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Eye pain (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Feces discolored (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Obsessive thoughts (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No